CLINICAL TRIAL: NCT02897674
Title: The Chemical Structure of a Lipid Determines Its Effect on Blood Lipid Profile and Fat Deposition
Brief Title: Effect of Palm Olein Intake on Lipid Profile and Fat Deposition
Acronym: PalmOil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15HH2616
Record Dates: First submitted 2016-08-17; First posted 2016-09-13 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: palm oil; lipid profile
MeSH Terms: interventions — Soybean Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight (Experimental): Participants will BMI 18.5-24.9 kg/m2 will consume 20% of their calories from one of the three dietary fats Intervention: palm olei Intervention: interesterified palm olein Intervention: soybean oil
  Interventions: Dietary Supplement: Palm olein; Dietary Supplement: Interesterified palm olein; Dietary Supplement: soybean oil
- Overweight (Experimental): Participants will BMI 25-29.9 kg/m2 will consume 20% of their calories from one of the three dietary fats Intervention: palm olei Intervention: interesterified palm olein Intervention: soybean oil
  Interventions: Dietary Supplement: Palm olein; Dietary Supplement: Interesterified palm olein; Dietary Supplement: soybean oil

INTERVENTIONS:
Dietary Supplement: Palm olein — two thirds of the 30% fat calories will come from palm olein
Dietary Supplement: Interesterified palm olein — two thirds of the 30% fat calories will come from interesterified palm olein
Dietary Supplement: soybean oil — two thirds of the 30% fat calories will come from soybean oil

SUMMARY:
Aims: To investigate whether diet with realistic doses on palm oil will have an effect on lipid profile and fat deposition in healthy volunteers.

DETAILED DESCRIPTION:
Design: Randomized, parallel design over 14 weeks including a 2 week standardization period and 12 week supplementation. In the standardization period all participants will incorporate palm oil into their diet which will make up 20% of their calories providing a baseline measure. In the supplementation period of 12 weeks, each volunteer will be randomized into one of the three fats: palm olein, interesterified palm olein or soybean oil, consuming 20% of their calories from these fast and remaining 10% fat calories from fats naturally occurring in foods like meat and nuts. Otherwise participants will keep the rest of their diet habitual.

Population: 60 healthy males and females aged between 18 and 60 years, of which 30 participants with a BMI between 18.5-24.9kg/m2 and 30 participants with a BMI between 25-29.9kg/m2 and fasting plasma glucose and no evidence of insulin resistance will be recruited. No pre-existing morbidity including cardiac, hepatic or renal disease, history of diabetes, hypertension or hyperlipidemia.

Treatment: Pre-intervention: Participants will be asked to record habitual dietary intake by completion of a 4-day food diary and be asked to wear an accelerometer armband to assess physical activity at the beginning and at the end of supplementation period.

2 weeks standardization period: All participants will be asked to replace added fat in their diet with palm olein providing two thirds of 30% fat calories.

At the end of the standardization period, which will be the first day of a 12 week dietary intervention, as well as at the end of 12 week supplementation, participants will attend the clinical research facility for a study visit. Weight, height and waist circumference will be taken; total and regional body composition will be measured by MRI. Fasting and post prandial plasma glucose, insulin, appetite hormones and lipids will be measured. Participants will be asked to come in for follow-up visits at week 6 and 10 for a single blood samples and weight check.

12 week supplementation period: participants will be randomized into one of the three supplementation groups: palm olein, interesterified palm olein or soybean oil. Participants will be asked to consume two thirds of their 30%fat calories from one of the oils while incorporating it into their normal diet in cooking and baking.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: 30 healthy volunteers (male and female), of all ethnicities, aged 18-60 years, with a body mass index (BMI) of 18.5-25kg/m2.
* Phase II: 30 healthy volunteers (male and female), of all ethnicities, aged 18-60 years, with a BMI of 25-29.9kg/m2.

Exclusion Criteria:

* Following a high fat diet (more than 40% calories coming from fat)
* Abnormal liver function test (elevated alanine aminotransferase and aspartate transaminase)/ abnormal kidney function test (elevated plasma creatinine)
* History of type 2 diabetes mellitus, cancer, stomach ulcers, drug abuse or alcoholism, gastrointestinal disorders like Crohn's disease
* Smokers
* On lipid/blood pressure- lowering medication/supplements
* Blood pressure>140/90 mm Hg
* Fasting total cholesterol > 6.2 mmol/L
* Fasting triacylglyceride > 2.0 mmol/L
* Candidates who are going abroad during the planned schedule for the dietary intervention
* Subject must not be allergic to intervention
* Pregnancy and breastfeeding (pregnancy test will be undertaken at the screening visit)
* Subjects taking nutritional supplements or on any weight-loss programs
* Subjects who gained or lost ≥ 3kg weight in the past three months
* Female subjects were not on oral contraceptives.
* Subjects with history of hypo- and hyperthyroidism
* Claustrophobia
* Metal implants for example cardiac pacemakers and join replacement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total cholesterol following the supplementation | fasting measure in week 3, 6, 10, 14

SECONDARY OUTCOMES:
Change from baseline in body composition | Fasting measure in week 3 and week 14
  total and regional body composition assessed by MRI
Change from baseline in lipoproteins | time=0 in week 3, 6, 10, 14
Postprandial change in appetite hormones | time=-15, -5,15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, 480 in week 3 and week 14

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Research Facility — http://imperial.crf.nihr.ac.uk/